CLINICAL TRIAL: NCT02270034
Title: Phase Ib, Open-label, Multicenter, Dose-escalation Study Followed by an Extension Phase to Evaluate the Safety and Activity of the Combination of Crizotinib With Temozolomide and Radiotherapy in Patients With Newly Diagnosed Glioblastoma
Brief Title: Study to Evaluate Safety and Activity of Crizotinib With Temozolomide and Radiotherapy in Newly Diagnosed Glioblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Grupo Español de Investigación en Neurooncología (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEINO 1402
Record Dates: First submitted 2014-10-14; First posted 2014-10-21 (Estimated); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: Glioblastoma Multiforme (Grade IV) of Cerebellum
MeSH Terms: conditions — Glioblastoma | interventions — Crizotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cohort crizotinib (Experimental): Combination of crizotinib with temozolomide and radiotherapy following Stupp regime
  Interventions: Drug: Crizotinib

INTERVENTIONS:
Drug: Crizotinib — Crizotinib is added to Stupp method

SUMMARY:
This multicenter, open-label, phase Ib trial aims to assess the safety and activity and safety of crizotinib (in combination with radiotherapy and temozolomide) in adult patients with newly diagnosed glioblastoma.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and the willingness to sign a written informed consent document.
2. Male or Female ≥18 years old and ≤ 70 years old
3. Newly diagnosed glioblastoma (GB) confirmed by biopsy or resection 4-7 weeks before registration.
4. Patients must have at least 15 unstained slides or 1 tissue block (frozen or paraffin embedded) available from a prior biopsy or surgery (archival tumor material).
5. Patients must have sufficient time for recovery from prior surgery (at least 4 weeks).
6. Karnofsky Performance Score (KPS) ≥ 60%.
7. Adequate hematologic function: Hemoglobin ≥ 10 g/dL, Leukocytes > 3,000/mcL, absolute neutrophil count (UNL) ≥ 1,500 cells/ul, platelets ≥ 100,000 cells/ul.
8. Adequate liver function: Bilirubin ≤ 2 X upper limit of normal (ULN); aspartate aminotrasferase (AST) (SGOT) ≤ 2.5 X ULN
9. Creatinine within normal institutional limits or creatinine clearance > 60 mL/min/1.73 m2l for subjects with creatinine levels above institutional normal.
10. The effects of crizotinib on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or harrier method of birth control; abstinence; surgical sterilization) prior to study entry and for the duration of study participation and for at least 3 months thereafter. The definition of effective contraception will be based on the judgment of the principal investigator or a designated associate. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. All female patients with reproductive potential must have a negative pregnancy test (serum/urine) within 2 weeks prior to starting treatment.

Exclusion Criteria:

1. Presence of extra-cranial metastatic disease.
2. Any prior radiotherapy (RT) or chemotheraphy (QT) treatment.
3. Patients must not have received prior Gliadel wafers.
4. The use of enzyme-inducing antiepileptic drugs will not be allowed. Those patients taking enzyme-inducing antiepileptic drugs required a 7-day washout period before registration.
5. Any surgery (not including minor diagnostic procedures such as lymph node biopsy) within 2 weeks of baseline disease assessments; or not fully recovered from any side effects of previous procedures.
6. Any clinically significant gastrointestinal abnormalities, which may impair intake, transit or absorption of the study drug, such as the inability to take oral medication in tablet form.
7. Any psychiatric or cognitive disorder that would limit the understanding or rendering of informed consent and/or compromise compliance with the requirements of this protocol.
8. Uncontrolled or significant cardiovascular disease, including:

   * A myocardial infarction within 12 months;
   * Uncontrolled angina within 6 months;
   * Congestive heart failure within 6 months;
   * Diagnosed or suspected congenital long QT syndrome;
   * Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes);
   * Prolonged corrected QT (QTc) interval on pre-entry electrocardiogram (>470 msec);
   * Any history of second or third degree heart block (may be eligible if currently have a pacemaker);
   * Heart rate <50/minute on pre-entry electrocardiogram;
   * Uncontrolled hypertension.
9. Any patient with a history of significant cardiovascular disease, even if currently controlled, or who has signs or symptoms suggesting impaired left ventricular function in the judgment of the investigator must have a screening left ventricular ejection fraction (LVEF) evaluation by ECHO or angyography (MUGA). Patients with LVEF measurements below local institutional lower limit of normal or less than 50% will not be eligible.
10. Individuals with a history of a different malignancy are ineligible except for the following circumstances: Individuals with a history of other malignancies are eligible if they have been disease-free for at least 3 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 3 years: cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin. Patients will not be eligible if they have evidence of other malignancy requiring therapy other than surgery within the last 3 years.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-08-13 (Actual); Primary Completion 2020-10-26 (Actual); Study Completion 2020-10-26 (Actual)

PRIMARY OUTCOMES:
Treatment safety | 7 months
  Number of participants with adverse events as a measure of safety and tolerability

SECONDARY OUTCOMES:
Recommended dose in phase II | 7 months
  Based on pharmakinetic analysis by Cmax
Anti-tumor activity | 7 months
Overall Survival | Two years
  Time between start of treatment and death

CONTACTS AND LOCATIONS:
Overall Officials: Juan Manuel Sepúlveda, MD, Study Chair — Hospital 12 de Octubre; María Martínez, MD, Study Chair — Hospital del Mar
Locations (4):
- Spain (4):
  - Institut Català D'Oncologia L'Hospitalet (Ico), L'Hospitalet de Llobregat, Barcelona
  - Hospital Del Mar, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid